CLINICAL TRIAL: NCT01434849
Title: Phase 1 Study of Topical Beta Blocker to Prevent the Proliferative Stage of Infantile Hemangioma
Brief Title: Timolol for the Prevention of Proliferation of Infantile Hemangioma (TiPPIH Trial)
Acronym: TiPPIH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty with enrolled patients to complete trial.
Sponsor: Alice K. Gong (Other)
Responsible Party: Sponsor-Investigator, Alice K. Gong, Professor of Pediatrics, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSC20110333H
Record Dates: First submitted 2011-08-31; First posted 2011-09-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Infantile Hemangioma; Very Low Birth Weight Infants
Keywords: infantile hemangioma; very low birth weight infants; premature infants
MeSH Terms: conditions — Hemangioma, Capillary; Premature Birth | interventions — Timolol; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Timolol (Experimental): Application of 1-2 drops of Timolol maleate 0.5% ophthalmic aqueous solution to hemangioma twice daily.
  Interventions: Drug: topical 0.5% Timolol maleate
- Placebo (Placebo Comparator): Application of 1-2 drops of placebo gel twice daily to hemangioma.
  Interventions: Drug: Control (placebo) group

INTERVENTIONS:
Drug: topical 0.5% Timolol maleate — topical 0.5% Timolol aqueous solution, 1-2 drops to cover the hemangioma, twice daily
  Arms: Timolol
Drug: Control (placebo) group — Aqueous placebo, 1-2 drops to cover the hemangioma, twice daily
  Arms: Placebo

SUMMARY:
The purpose of this trial is to see if a topical beta blocker is effective in preventing the proliferation of infantile hemangioma.

DETAILED DESCRIPTION:
Infantile hemangiomas (IH) are among the most common, benign vascular tumors of infancy with an estimated prevalence of 4-5% of the population. IH are not found at birth but become evident within the first few weeks of life. They are characterized by a rapid proliferative phase that can last up to 4-6 months or longer and then a period of minimal or absent growth before an involutive phase where they may resolve with minimal or no scarring over multiple years. Although frequently thought of as benign lesions, hemangiomas can occur in locations to cause functional impairment of vital organs, can lead to ulcerations, scarring or disfigurement, and can lead to life-threatening complications. Management of these problematic IH includes laser, long-term systemic corticosteroids, interferon, Vincristine, surgery, and most recently systemic propranolol. Pulsed-dye laser is the only treatment approved by the FDA; it has been useful for superficial hemangiomas but has little effect on subcutaneous or deep-seated hemangiomas. The proposed therapeutic effects of propranolol are vasoconstriction, decreased expression of vascular endothelial growth factor (VEGR) and basic fibroblast growth factors (bFGF) genes through downregulation of Raf/mitogen-activated protein kinase pathway, and apoptosis of capillary endothelial cells. For periorbital lesions that may cause amblyopia or anisometropia, topical Timolol has been reported to be of benefit. There is one retrospective review that is proof of concept that shows that topical timolol is safe and effective treatment for 6 cases of IH.

The advantage of a topical therapy is the decreased risk of systemic side effects compared with oral or intravenous administration. The disadvantage is that limited penetration may preclude effectiveness for the thicker or deeper lesions.

Being of low birth weight as well as prematurity are known risk factors for IH. In the premature infant development clinic at the University of Texas Health Science Center in San Antonio infants less than 1500 grams birth weight are followed for three years following discharge from the Newborn Intensive Care Unit (NICU); approximately 16% of these infants have hemangiomas. Therefore the investigators find it reasonable to start treatment with a topical beta blocker at an early stage of hemangioma to prevent the growth and proliferation and hence the possible severe effects associated with growth and thus impairment of vital organs/tissues.

ELIGIBILITY:
Inclusion Criteria:

* Babies admitted to NICU or seen in follow clinic that have a diagnosis of hemangioma that is verified by Principal Investigator (PI) or Co-Principal Investigators.

Exclusion Criteria:

* Babies with PHACES (Posterior fossa, Hemangioma, Arterial lesions, Cardiac abnormalities, Eye abnormalities) syndrome
* Babies with cardiac conditions that may predispose to heart block
* Babies with persistent hypoglycemia
* Babies on medications that may interact with beta blockers
* Babies who are hemodynamically unstable and are requiring pressors to maintain blood pressure
* Babies who are on systemic corticosteroid therapy

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2012-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in treatment group compared to placebo group with at least 50% improvement in the extent of hemangioma as compared to each other with respect to changes from baseline photographs. | 6 months
  hemangioma once detected will be measured and photographed. Measurements and photographs will be obtained every 2 weeks while the patient is in hospital and monthly after discharged until end point of 6 months.

SECONDARY OUTCOMES:
Compare treatment group to placebo group assessments | 6 months
  Difference in color of the hemangioma of the treatment group versus control group
Compare treatment group to placebo group assessments | 6 months
  More significant Retinopathy of Prematurity findings between treatment group versus control group
Compare treatment group to placebo group assessments | 6 months
  Frequency of adverse events (e.g. hypotension, behavioral changes, etc.) collected by investigator and reported by NICU staff and parents.

CONTACTS AND LOCATIONS:
Overall Officials: Alice K Gong, M.D., Principal Investigator — The University of Texas Health Science Center at San Antonio; Alice K Gong, MD, Study Director — University of Texas
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Many participants did not complete trial so there is not enough data to share.